CLINICAL TRIAL: NCT06389825
Title: Unravelling the Impact of Diet on Cardiovascular Health in Treated Heterozygous Familial Hypercholesterolemia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean-Philippe Drouin-Chartier, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FH-Diet-RX
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Familial Hypercholesterolemia; Nutrition, Healthy; Cholesterol, Elevated
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia | interventions — Diet, Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Canada's Food Guide principles (CFG diet) (Experimental): During 28 days, participants will receive de CFG diet. The CFG diet emphasizes low intakes of red and processed meats and high intakes of minimally processed plant foods with water as the drink of choice, as per Canada's Food Guide. The number of portions of protein foods, whole-grains, fruits and vegetables to be served daily reflects the recommended ¼-¼-½ proportions. Regarding protein quality, vegetable proteins are served more often than animal proteins as stated in Canada's Food Guide. Weekly, red meat is served once, two days are meatless, and one day is free of animal products.
  Interventions: Other: Healthy diet
- Standard North American diet (NAD diet) (Experimental): During 28 days, participants will receive de NAD diet. The NAD diet reflects current dietary intakes of the French-Canadian adult population in terms of foods, nutrients, and diet quality, as characterized in recent surveys conducted in an age- and a sex-representative sample of adults from the Province of Quebec. Intakes of minimally processed fruits and vegetables will be low; animal proteins, mostly red and processed meats, will be consumed more often than vegetable proteins; grains will be mostly refined; and ready-to-eat/ready-to-heat foods and sugary beverages will be served daily.
  Interventions: Other: Healthy diet

INTERVENTIONS:
Other: Healthy diet — 28-day fully controlled dietary intervention during which participants will receive a diet that reflects the recommendations of Canada's Food Guide.

SUMMARY:
The investigators will conduct a fully controlled dietary randomized crossover trial (RCT) including 10 adults with HeFH using lipid-lowering medication to investigate the impact of a diet low in red and processed meats and high in plant foods, reflecting Canada's Food Guide, in place of a standard North-American diet on LDL-cholesterol (LDL-C) levels and the plasma metabolome.

DETAILED DESCRIPTION:
The dietary intervention will be undertaken as a crossover RCT at the Institute on nutrition and functional foods (INAF, Laval University) in Quebec City. Participants (men and women with genetically-defined HeFH) will consume in a random order a fully-controlled diet low in red and processed meats and high in plant foods, reflecting Canada's Food Guide principles (CFG diet in further sections), and a standard North American diet (NAD diet; i.e. control diet), reflecting current dietary intakes of French-Canadians, for 4 weeks each, and separated by a 4-week washout period.

Once enrolled, participants will provide a blood sample and complete a self-administered, validated web-based food-frequency questionnaire. Participants will be randomly assigned to either the CFG-NAD or NAD-CFG diet sequence, using a computer-assisted program. The randomization (1:1) will be stratified by sex and LDL-receptor (LDLR) genotype. The two diets will be consumed for 4 weeks and separated by a 4-week washout period. During diet phases, all meals and foods will be provided to ensure optimal diet control using a 7-day cyclic menu. The CFG diet emphasizes low intakes of red and processed meats and high intakes of minimally processed plant foods with water as the drink of choice, as per Canada's Food Guide. The NAD diet reflects current dietary intakes of the French-Canadian adult population in terms of foods, nutrients, and diet quality, as characterized in recent surveys conducted in an age- and a sex-representative sample of adults from the Province of Quebec. An experienced food technician will prepare the diets. Each food and ingredient will be weighed with a precision of ±0.1 g.

On weekdays, subjects will visit INAF Clinical Research Unit to consume their lunch meal under the research coordinator's supervision. At that time, they will also be given their evening meals and the next day's packaged breakfast to take home. Weekend meals will be provided at the Friday visits. A checklist will be provided to all participants to identify the consumed foods.Alcohol, vitamin supplements, and natural health products will not be allowed. Tea and coffee (black) will be allowed (≤2 servings/day without daily fluctuations). Participants will be instructed to maintain their usual physical activity level. At the end of each diet, fasting plasma samples will be collected in ethylenediaminetetraacetic acid (EDTA) tubes. Parts of the samples will be stored at -80℃ for future ancillary analyses. Participants' anthropometry, body composition (DEXA scan), and blood pressure will be measured. To incorporate gender aspects associated with the intervention in knowledge transfer activities, subjects' appreciation of the diets will be assessed using visual analog scales filled after each meal on day 7 and 28 of each diet.

Objective 1: To investigate the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on LDL-C concentrations - the primary treatment target in HeFH management. This objective will output a convincing demonstration of the cholesterol-lowering effects of diet in adults with HeFH, supporting the effectiveness of dietary interventions in HeFH management. Investigators will compare post-diet LDL-C levels (primary outcome) using mixed models for repeated measures. Secondary outcomes include other atherogenic lipoproteins and lipids (apolipoprotein B, non-HDL-C, total-C, triglycerides, lipoprotein (a)) and other cardiovascular disease risk factors (fasting plasma glucose, fasting insulin, systolic and diastolic blood pressure, FH risk score, 10-year risk of cardiovascular disease). Potential effect modification by key participant characteristics (age, BMI, sex, LDLR genotype, lipoprotein (a) and diet sequence) will also be tested.

Objective 2: To assess the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on the plasma metabolome. This objective serves a dual purpose as it will: 1. inform on the dietary impact on systemic metabolism, beyond its impact on LDL-C levels, further supporting the importance of healthy dietary habits in HeFH; and 2. allow the identification of an unbiased HeFH-specific plasma metabolomic signature of a diet low in red and processed meats and high in plant foods to be used as an objective proxy of diet adherence. To document post-diet differences in plasma metabolome and identify the metabolomic signature of the CFG diet, investigators will derive a reproducible multi-metabolite model discriminating the post-CFG/post-NAD metabolomic profiles.

Results will fill key gaps on the short- and long-term influence of diet on cardiovascular health in HeFH.

ELIGIBILITY:
Inclusion Criteria:

* Genetically-defined HeFH
* Premenopausal women with a regular menstrual cycle for >3 months
* Postmenopausal women (without hormone replacement)

Exclusion Criteria:

* Age >60 years
* Homozygous FH
* Personal history of cardiovascular disease
* Prevalent diabetes or anti-diabetic drug use
* Severe obesity
* Unstable body weight for >3 months
* Uncontrolled hypertension
* Genetic hypertriglyceridemia
* Allergies/aversions to components of the experimental diets
* Any other condition that would interfere with optimal participation in the intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Post-diet differences in LDL-cholesterol concentrations. | This analysis will compare LDL-C levels from plasma samples collected at the end (day 28) of each diet
  Investigators will evaluate the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on LDL-cholesterol concentrations among 10 adults with HeFH.

SECONDARY OUTCOMES:
Post-diet differences in other atherogenic lipoproteins and lipids | This analysis will compare levels of atherogenic lipoproteins and lipids measured from plasma samples collected at the end (day 28) of each diet
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on plasma levels of atherogenic lipoproteins and lipids (apolipoprotein B, non-HDL-cholesterol, total-cholesterol, triglycerides, lipoprotein(a)).
Post-diet differences in C-reactive protein levels | This analysis will compare C-reactive protein levels (mg/L) measured at the end (day 28) of each diet.
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on C-reactive protein levels (mg/L).
Post-diet differences in systolic and diastolic blood pressure | This analysis will compare systolic and diastolic blood pressure (mm Hg) measured at the end (day 28) of each diet.
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on systolic and diastolic blood pressure (mm Hg).
Post-diet differences in 10-year risk of atherosclerotic cardiovascular disease | This analysis will compare 10-year risk of atherosclerotic cardiovascular disease (%) measured at the end (day 28) of each diet.
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on 10-year risk of atherosclerotic cardiovascular disease (%).
Post-diet differences in plasma metabolomics profiles | This analysis will compare metabolomic profiles from plasma samples collected at the end (day 28) of each diet.
  Investigators will assess the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on the plasma metabolome among 10 adults with HeFH. Plasma metabolites will be measured using 3 complementary liquid chromatography-tandem mass spectroscopy methods for 1) polar metabolites (e.g. amino acids), 2) lipids, and 3) free fatty acids. Relative abundance of the metabolites will be compared between the two diets.

OTHER OUTCOMES:
Post-diet differences in appetite sensation | Appetite sensation was measured at the end of the first (day 7) and the last week (day 28) of each diet. Changes between day 28 and day 7 will be calculated and compared between diet.
  Investigators will compare between-diet changes in appetite sensation between the first and the last week of each diet in a gender specific approach. Appetite sensation was measured using visual analog scale at the end of the first (day 7) and the last week (day 28) of each diet. Changes between day 28 and day 7 will be calculated and compared between diet.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Drouin-Chartier, PhD, Principal Investigator — Laval University
Locations (1):
- INAF-NUTRISS Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided